CLINICAL TRIAL: NCT01881555
Title: FUnctional Testing Underlying Coronary REvascularisation.
Acronym: FUTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.725; Numéro ID RCB : 2012-A01195-38 (Other: ANSM)
Record Dates: First submitted 2013-05-29; First posted 2013-06-19 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2018-06

CONDITIONS: Multivessel Coronary Artery Disease; Vessel Disease; Stable Angina; Unstable Angina or Stabilized Non-ST Elevated Myocardial Infarction; Patients With ST-elevated Myocardial Infarction; Revascularization of Culprit Coronary Artery
Keywords: fractional flow reserve; multivessel coronary artery disease; angiography
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FRACTIONAL FLOW RESERVE (Other): Patients will have FFR measured in each diseased vessel identified by the coronary angiographic evaluation. Intra-coronary adenosine (at least 100 micrograms performed 2 times) OR intravenous adenosine (at a dose of 140µg/kg/min during at least 4 minutes) will be administered prior to FFR assessment.
  Revascularization strategy will be based upon FFR findings and revascularization either by coronary stenting or CABG will only be performed on target lesions with FFR≤0.8.
  Interventions: Procedure: invasive coronary angiography
- ANGIOGRAPHY (Other): Patients undergo an angiography. Based on angiographic evaluation, the physicians define the revascularization strategy.
  Interventions: Procedure: Functional testing by fractional flow reserve measurement

INTERVENTIONS:
Procedure: invasive coronary angiography
  Arms: FRACTIONAL FLOW RESERVE
Procedure: Functional testing by fractional flow reserve measurement — Functional testing by fractional flow reserve measurement
  Arms: ANGIOGRAPHY

SUMMARY:
The objective of this trial is to compare the clinical outcomes and cost-effectiveness of 2 therapeutic strategies, one based on coronary angiography guidance and the other based on coronary angiography with fractional flow reserve (FFR) in multivessel coronary artery disease patients.

The trial is a prospective, multicenter, French, randomized clinical trial including men and women ≥ 18 years presenting with significant multivessel disease defined by coronary angiography as coronary narrowing > 50% diameter stenosis in at least 2 major epicardic vessels. The patients who give their informed consent will be randomly assigned to a therapeutic strategy based upon coronary angiography or angiography with FFR testing. In the FFR group, a significant coronary stenosis will be defined by a FFR ≤ 0.8. Based upon this multivessel evaluation (angiography or FFR), the investigator will choose the best therapeutic strategy to his discretion (medical optimal treatment, coronary stenting, coronary artery bypass graft surgery). The aim of revascularization procedures will be to obtain complete revascularization. In the FFR group, only stenosis with FFR≤0.8 will be treated.

The primary end point of the trial is a composite of major cardiovascular events including death from any cause, myocardial infarction, any hospitalization for coronary revascularization performed in addition to initial treatment and stroke at 1 year of follow-up.

Secondary end points will include adverse events, individual major cardiovascular events, stent thrombosis, bleeding events, occlusion of coronary artery bypass graft, patient's quality of life and cost-effectiveness and 30-day, 6 month, 2-year and 5-year outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* referred to the cardiologist for one of the following medical condition :

  * ST segment elevation myocardial infarction evolving for more than 7 days after revascularization of culprit coronary artery or
  * no ST elevation acute coronary syndrome with or without troponin (T or I) elevation and medically stabilized for at least 12 hours or
  * stable angina (CCS I, II or III) or
  * chest pain diagnosis with suspicion of CAD or with ischemia certificated by non invasive tests.
  * patients with at least 2 vessel disease (≥50% stenosis on angiography) including the left anterior descending coronary artery or with single vessel disease on left main coronary artery
* Patient willing and able to provide informed, written consent
* Patient not under legal protection
* Patient benefiting from the French Health Insurance

Exclusion Criteria:

* Pregnancy, childbearing, absence of effective contraception
* Previous coronary bypass surgery
* Planned associated valvular surgery
* Life expectancy < 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2013-05-27; Primary Completion 2017-06-10 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
composite endpoint that includes the rate of major cardiovascular events defined as a composite of death from any cause, myocardial infarction, any hospitalization leading to additional coronary revascularization, stroke. | 1 year.
  The effect of therapeutic strategy will be assessed by the reduction of the incidence of major cardiovascular events in the group "angiography with FFR testing" in comparison to the group "angiography alone". Patients will be prospectively and clinically followed during the duration of the study and all major cardiovascular events will be documented and reported in the electronic case report form.
Bypass graft patency assessed in all CABG patients at one year by coronary multidetector computed tomography . | 1 year

SECONDARY OUTCOMES:
Major cardiovascular events in all patients, in diabetic patients, by revascularization strategy (angioplasty, coronary artery bypass graft surgery, medical optimal treatment). | 1 year
The effect of our therapeutic strategy will be assessed upon each category of cardiovascular event individually. | 1 year
Major cardiovascular events in all patients. | 2 years, 3 years, 4 years and 5 years
Stent thrombosis. | 1 year
Bleeding events. | 1 year
Patient's quality of life | 1 year
  We will use the European Quality of Life-5 Dimensions instrument.
Cost-effectiveness of each therapeutic strategy | 1 year
  NACost-effectiveness of each therapeutic strategy will be assessed by the evaluation of medical costs linked to the pathology (hospitalizations, consultations, and external medical costs (biology, radiology, medications) and compared in the 2 groups during the first 12 months of follow up.
Bypass graft patency assessed in all CABG patients at one year by coronary multidetector computed tomography . | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- HOSPICES, Lyon, France

REFERENCES:
- [Result] Rioufol G, Derimay F, Roubille F, Perret T, Motreff P, Angoulvant D, Cottin Y, Meunier L, Cetran L, Cayla G, Harbaoui B, Wiedemann JY, Van Belle E, Pouillot C, Noirclerc N, Morelle JF, Soto FX, Caussin C, Bertrand B, Lefevre T, Dupouy P, Lesault PF, Albert F, Barthelemy O, Koning R, Leborgne L, Barnay P, Chapon P, Armero S, Lafont A, Piot C, Amaz C, Vaz B, Benyahya L, Varillon Y, Ovize M, Mewton N, Finet G; FUTURE Trial Investigators. Fractional Flow Reserve to Guide Treatment of Patients With Multivessel Coronary Artery Disease. J Am Coll Cardiol. 2021 Nov 9;78(19):1875-1885. doi: 10.1016/j.jacc.2021.08.061. PMID 34736563